CLINICAL TRIAL: NCT04093622
Title: Long-term Follow-Up Study Following Treatment With Fate Therapeutics' Engineered Cellular Immunotherapy
Status: Terminated | Type: Observational
Why Stopped: Incorporation of LTFU into the main interventional study.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: FT-004
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2021-12

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Multiple samples including: whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genetically engineered NK Cell - treated: Long term follow-up of subjects who have received lentivirus-mediated genetically engineered NK Cells.
  Interventions: Genetic: Genetically engineered NK cells

INTERVENTIONS:
Genetic: Genetically engineered NK cells — No study drug is administered in this study. Subjects who received lentivirus-mediated genetically engineered NK Cells in a previous trial will be evaluated in this trial for long-term safety and efficacy.

SUMMARY:
The purpose of the study is to assess long-term side effects from subjects who receive a Fate Therapeutics genetically modified NK cell product. Subjects who previously took part in a Fate Therapeutics study and received genetically changed NK cells will take part in this long-term follow-up study. Subjects will join this study once they complete the parent interventional study. No additional study drug will be given, but subjects can receive other therapies for their cancer while they are being followed for long term safety in this study.

For a period of 15 years starting from the last administration of Fate Therapeutics genetically modified NK cell product, subjects will be assessed for long-term safety and survival through questionnaires and blood tests.

DETAILED DESCRIPTION:
This is a non-therapeutic, multi-center, long-term follow-up (LTFU) study of subjects who received a Fate Therapeutics NK cell product that has been modified by lentivirus-mediated genetically engineering. The period of follow-up is 15 years after the administration of the NK cell product.

The study involves up to 15 years post-infusion monitoring of subjects who have been exposed to lentivirus-mediated gene transfer in Fate Therapeutics clinical studies. Upon withdrawal or completion of the parent interventional study, the study site will contact the subject/healthcare provider/legal guardian annually.

ELIGIBILITY:
Inclusion Criteria:

* Received engineered cellular immunotherapy in a Fate Therapeutics Interventional Study

Exclusion Criteria:

• Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects hematological malignancies rolling over from interventional study where they were treated with Fate Therapeutics genetically modified NK cell product.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) post-infusion | 15 years post last treatment
  OS defined as the interval between the date of first Fate Therapeutics genetically modified NK cell product infusion and date of death due to any cause.

SECONDARY OUTCOMES:
Incidence of LTFU adverse events (AEs), including serious adverse events (SAEs) associated with administration of Fate Therapeutics genetically modified NK cell product that have been genetically modified by lentiviral vectors. | 15 years post last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Elstrom, MD, Study Director — Fate Therapeutics
Locations (5):
- United States (5):
  - Mayo Clinic, Phoenix, Arizona
  - UC San Diego, San Diego, California
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No